CLINICAL TRIAL: NCT02388256
Title: Acupuncture for Enhanced Recovery After Surgery in Patients Undergoing Laparoscopic Colorectal Cancer Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korean Medicine Hospital of Pusan National University (Other)
Responsible Party: Principal Investigator, Gyung-Mo Son, Associate professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 03-2014-012
Record Dates: First submitted 2015-03-01; First posted 2015-03-13 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Colorectal Cancer
Keywords: colon; colorectal; cancer; neoplasm
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): Manual and electroacupuncture
  Interventions: Device: acupuncture
- Enhanced recovery program after surgery (Active Comparator): Enhanced recovery program after surgery
  Interventions: Device: acupuncture; Other: early recovery program after surgery

INTERVENTIONS:
Device: acupuncture — Points of Stomach 36 (ST36), Stomach 37 (ST37), Liver 3 (LR3), Large Intestine 11 (LI11), Large Intestine 4 (LI4), Spleen 6 (SP6), Spleen 4 (SP4) and Pericardium 6 (PC6) will be used. Electrical stimulation with alternating frequency of 2 to 100 Hz will be applied to the selected points (LI4 to LI11, ST36 to ST37, and bilateral SP6).
  Rationale of acupuncture treatments will include both traditional theory of harmonizing gastrointestinal function and strengthening vital energy as well as modern experimental and clinical evidence of regulating gastrointestinal motility and other symptom managements. Treatments will be provided by qualified hospital staff (Korean medical doctors) with more than 10 years of clinical experience.
Other: early recovery program after surgery — An enhanced recovery program after surgery that was designed and is currently implemented by surgeons, anesthetists, dietitians, and nurses will be provided. The program includes preoperative education, early water/food intake, early mobilization, early removal of Foley catheter and drains, structured nursing care, and nutritional support.
  Other Names: fast-track recovery program
  Arms: Enhanced recovery program after surgery

SUMMARY:
Background:

Patients who undergo laparoscopic surgical resection of colorectal cancer may experience various post-operative symptoms (e.g., pain, nausea and vomiting, and anxiety) and limitation of daily activities (e.g., walking capacity). There is also a risk of post-operative complications and a prolonged hospital stay due to complications. Patients who underwent surgical resection may have experienced chronic pain, anxiety/depression, or diminished quality of life. The physical, psychological, and functional aspects of patients' disorders imply the necessity of multidisciplinary care, including complementary or traditional medicines such as acupuncture. This study aims to assess whether acupuncture treatment, combined with an enhanced recovery program after surgery in an inpatient care setting is effective than only an enhanced recovery program after surgery.

Objective:

To assess the effectiveness and safety of acupuncture combined with an enhanced recovery program after surgery to reduce postoperative symptoms and improve functional recovery and the patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparoscopic surgery of colorectal cancer resection (right hemicolectomy, left hemicolectomy, anterior resection with primary anastomosis, and low anterior resection with loop ileostomy for fecal diversion)
* Patients aged 18 to 75
* American Society of Anesthesiologists Grade 1 to 2
* Eastern Cooperative Oncology Group Grade 0 to 2
* Written informed consents

Exclusion Criteria:

* Pregnancy
* Inflammatory bowel disease
* Comorbidities that may affect outcomes of surgery (e.g., chronic kidney disease, chronic liver disease, cardiopulmonary failure, and diabetes with complications)
* Resection of other organs for radical removal of colorectal cancer
* Patients requiring enterolysis due to previous history of abdominal surgery
* Obstructive colorectal cancer
* Metastatic colorectal cancer
* Cognitive impairment that may affect the patient's ability to complete the outcome assessments
* Previous history of stroke
* Previous history of sensitive reaction to acupuncture
* Patients unable to cooperate with acupuncture treatments
* Pacemaker implantation
* Previous history of epilepsy
* Patients who have received Korean medicine treatments (acupuncture, moxibustion, cupping, or herbal medicine) within 2 weeks
* Patients who have participated in other trials within 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Recovery of physical function | at 2 weeks after surgery
  Recovery of physical function, as measured by the physical function domain of European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) C30 instrument

SECONDARY OUTCOMES:
Pain intensity | at 4, 12, 24, 48, 72 hours after surgery, at 1 week after surgery (an expected day of discharge), at 2 weeks after surgery, and at 4 weeks after surgery
  Pain scores on a numeric rating scale. Score ranges from 0 (no pain at all) to 10 (the worst pain imaginable)
Time to first flatus | up to 1 week after surgery (an expected period of admission)
  elapsed time after surgery
Time to tolerate soft diet | up to 1 week after surgery (an expected period of admission)
  elapsed time after surgery
Time to first defecation | up to 1 week after surgery (an expected period of admission)
  elapsed time after surgery
Time to independent walk | up to 1 week after surgery (an expected period of admission)
  elapsed time after surgery
Number of insertions of nasogastric tube | up to 1 week after surgery (an expected period of admission)
  number of insertions of nasogastric tube
Incidence of nausea/vomiting | up to 1 week after surgery (an expected period of admission)
  number of nausea / vomiting reported by the patients
Time to first removal of Foley catheter | up to 1 week after surgery (an expected period of admission)
  elapsed time after surgery
Number of reinsertions of Foley catheter | up to 1 week after surgery (an expected period of admission)
  number of reinsertions of Foley catheter
Number of clean intermittent catheterizations | up to 1 week after surgery (an expected period of admission)
  number of clean intermittent catheterizations
Quality of life measured by EORTC QLQ C30 | at 2 weeks after surgery, at 4 weeks after surgery, and at 12 weeks after surgery
  Quality of life measured by EORTC QLQ C30
Patient's global assessment after surgery | at 4 weeks after surgery, at 12 weeks after surgery
  Response options include very much improved, somewhat improved, no change, somewhat worsened, and very much worsened.
Use of medication | at 1 week after surgery (an expected day of discharge), at 2 weeks after surgery, at 4 weeks after surgery, and at 12 weeks after surgery
  Use of analgesics, antiemetics and other medications after surgery
Anxiety and depression | at 2 weeks after surgery, at 4 weeks after surgery, at 12 weeks after surgery
  Patients' anxiety and depression level measured by the Hospital Anxiety-Depression Scale
Postoperative complications | within 12 weeks after surgery
  * wound infection
  * urinary tract infection
  * urinary retention
  * chest infection
  * other infection
  * paralytic ileus
Serious adverse events | within 12 weeks after surgery
  * respiratory failure requiring ventilation
  * renal failure requiring dialysis
  * cardiac failure
  * myocardial infarction
  * anastomotic leakage requiring surgery
  * anastomotic leakage requiring drainage
  * bowel obstruction/stricture requiring surgery
  * abdominal wall dehiscence requiring surgery
  * readmission within 30 days after surgery
  * reoperation within 30 days after surgery
  * mortality during surgery or within 30 days after surgery
Adverse events related to acupuncture | within 12 weeks after surgery
  Expected or unexpected adverse events that are considered to be associated with acupuncture treatments.

OTHER OUTCOMES:
Adherence to enhanced recovery program after surgery | at 1 week after surgery (an expected day of discharge)
  Number of patients who discharge the hospital at the expected day as planned

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Mo Son, PhD, Principal Investigator — Pusan National University Yangsan Hospital; Gi Young Yang, PhD, Principal Investigator — Korean Medicine Hospital, Pusan National University
Locations (2):
- South Korea (2):
  - National Clinical Research Centre for Korean Medicine, Korean Medicine Hospital, Pusan National University, Yangsan, Kyung Sang South Province
  - Pusan National University Yangsan Hospital, Yangsan, Kyung Sang South Province